CLINICAL TRIAL: NCT00809666
Title: A Prospective Randomised Study of Automated Versus Mercury Blood Pressure Recordings in Pregnancy
Brief Title: Measuring Blood Pressure in Pregnancy Using Mercury and Automated Device
Acronym: PRAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George Hospital, Australia (Other)
Responsible Party: Professor Mark Brown, St George Hospital and UNSW
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 00/41 Brown
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension; Pregnancy; Pre Eclampsia
Keywords: pregnancy; hypertension; mercury sphygmomanometry; blood pressure; automated blood pressure; pre eclampsia; Hypertension in pregnancy
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mercury (No Intervention): All subsequent blood pressure recording done using mercury sphygmomanometry
  Interventions: Device: Automated blood pressure recording device Omron HEM 705CP

INTERVENTIONS:
Device: Automated blood pressure recording device Omron HEM 705CP — All subsequent blood pressure recordings done using the automated device

SUMMARY:
The aim of the PRAM study was to determine whether women diagnosed with hypertension in pregnancy, using the traditional mercury device, have the same pregnancy outcomes when blood pressure is measured by either an automated device or a mercury device throughout the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women with a diagnosis of hypertension in pregnancy

Exclusion Criteria:

* non-pregnant and normotensive pregnancy women

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2000-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary maternal outcome measure was the number of women having any episode of severe hypertension (BP ³ 170/110mmHg).

SECONDARY OUTCOMES:
Secondary end points included gestation at birth, caesarean section and induction of labour rates.

CONTACTS AND LOCATIONS:
Locations (1):
- St George Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] High blood pressure research Council of Australia. Position Statement on the replacement of mercury sphygmomanometers. September 2006. www.hbprca.com.au
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394